CLINICAL TRIAL: NCT07118280
Title: Saliva Composition in Oculo-Pharyngeal Muscular Dystrophy (OPMD)
Brief Title: Oral Health, Saliva Viscosity and Composition in Oculo-Pharyngeal Muscular Dystrophy (OPMD)
Status: Recruiting | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-22-9824-AZ-CTIL
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Oculopharyngeal Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Oculopharyngeal

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Unstimulated whole saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with OPMD
- Control: Unaffected spouse or household member without OPMD

SUMMARY:
The goal of this observational study is to explore whether oral health and saliva viscosity and composition in Oculopharyngeal Muscular Dystrophy (OPMD) is different from control subjects.

The main questions it aims to answer are:

Do swallowing disturbances in OPMD adversely affect oral health? Is saliva thickness (viscosity) is increased in OPMD? Does saliva in OPMD contains biochemical markers of the disease?

DETAILED DESCRIPTION:
The objectives of this observational study is to investigate oral health, saliva rheology and explore biochemical markers in OPMD. specifically to determine if anecdotal reports of "thick saliva" represent a previously unrecognized manifestation of the disease.

Oculo-pharyngeal muscular dystrophy (OPMD) is a rare, late-onset, hereditary (OMIM 164300) progressive degenerative muscle disease characterized by oro-pharyngeal dysphagia and eyelid ptosis and skeletal muscle weakness.

Oro-pharyngeal dysphagia is associated with impaired oral health in elderly patients in general, in patients with neurodegenerative diseases and in Parkinson's disease. Yet, oral health in OPMD has not been explored so far. Additionally, a notion in one report that more than half of patients with OPMD complained about "having thick saliva" has not triggered further research of saliva properties in OPMD.

OPMD patients enrolled in IsrOPMD registry at the multidisciplinary OPMD service at the Sheba Medical Center will be offered to participate in the study. Unaffected spouse or household member of each patient will be offered to serve as a control. Subjects younger than 18 years of age and those with any condition that may affect a composition of saliva were excluded from this study.

All study subjects will proceed a thorough stomatological examination documenting the number of decayed, missing and filled teeth (DMFT index), dryness of oral mucosa, presence of tongue coating, atrophic papillae, cleft or geographic tongue, gingival inflammation and gross saliva secretion, unstimulated whole saliva flow rate and saliva viscosity. Untargeted metabolomic analysis of the saliva will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with OPMD and their spouses or household members

Exclusion Criteria:

* • Pregnancy or presence of any disease that may affect a composition of saliva

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Patients group: consisted OPMD patients enrolled in IsrOPMD registry at the multidisciplinary OPMD service at the Sheba Medical Center. The Control group: patients' spouse or household member without OPMD.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Saliva Viscosity | Upon enrollment in the study
  Viscosity of unstimulated whole saliva

SECONDARY OUTCOMES:
Oral health indices | Upon enrollment in the study
  DMFT, presence of tongue coating, clinical appearance of saliva and saliva-related complains

OTHER OUTCOMES:
Concentration of Metabolites in saliva | Upon enrollment in the study
  Differences in concentration of metabolites in unstimulated whole saliva of patients and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel